CLINICAL TRIAL: NCT05482854
Title: ANRS 175 RHIVIERA-01: Assessment of HIV Remission Upon Combination Antiretroviral Therapy (cART) Interruption in Early Treated Individuals From ANRS CO6 PRIMO Cohort Carrying the Major Histocompatibility Complex (MHC) B35/53Bw4TTC2 Genotype
Brief Title: Assessment of HIV Remission Upon cART Interruption in Early Treated Individuals Carrying the MHC B35/53Bw4TTC2 Genotype
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ANRS 175 RHIVIERA-01
Record Dates: First submitted 2022-01-03; First posted 2022-08-01 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: HIV Infections
Keywords: treatment interruption; HIV remission; Post-treatment control; HLA-B35; Early treatment
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: The trial will be a pilot "proof of concept", one arm, multicenter, nested in the ANRS CO6 PRIMO Cohort, in which the intervention is treatment interruption (of at least 6 months).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated early and carrying the MHC B35/53Bw4TTC2 Genotype (Experimental): Patients included in the ANRS CO6 PRIMO cohort, treated early and carrying the MHC B35/53Bw4TTC2 Genotype
  Interventions: Other: Analytical Treatment Interruption (ATI)

INTERVENTIONS:
Other: Analytical Treatment Interruption (ATI) — Analytical Interruption of Treatment for 24-48 weeks
  ART resumption and follow-up for 24 weeks if the participant meets at least one ART resumption criteria

SUMMARY:
The aim of the trial is to evaluate in ANRS CO6 PRIMO cohort participants if the presence of the MHC B35 (53) Bw4TTC2 genotype favors the control of HIV infection (defined by a viral load (VL) less than 400 cp/mL) after discontinuation of antiretroviral therapy (ART) initiated during primary HIV infection.

The trial will be a pilot "proof of concept", one arm, multicenter, nested in the ANRS CO6 PRIMO Cohort, in which the intervention is treatment interruption (of at least 6 months).

It is planned to include between 20 and 50 participants.

DETAILED DESCRIPTION:
The ANRS 175 RHIVIERA 01 trial will focus on people who were initiated early and have a particular genotypic profile associated with HIV remission.

The study proposes to test an intervention consisting in a ART-treatment interruption (of at least 6 months) in ANRS CO6 PRIMO cohort participants carrying the MHC B35/53Bw4TTC2 genotype and well controlled on cART.

The study aims to enrol 20-30 participants in 30 French clinical sites. Participants will be enrolled after checking eligibility criteria and will interrupt ART immediatly after inclusion.

Control of HIV-Infection, defined by a viral load less than 400 cp/mL, will be evaluated after 24 weeks of interruption.

Study duration will vary by participant, depending on the time of ART interruption and the time to viral rebound. Participants will be followed maximum 48 weeks on ATI. If there is a viral rebound justifying the resumption of ART, participant will be followed 24 weeks maximum after resumption. The maximum duration of the study will be 48+24 = 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years at the time of consent
* Enrolled and currently followed in a site of the ANRS CO6 PRIMO Cohort
* With the MHC genotype: at least one HLA B35 or B53 allele AND one HLA-A or B allele carrying the Bw4 epitope AND homozygous -21T residue in the HLA-B alleles AND heterozygous or homozygous for C2 epitope-carrying HLA-C alleles
* Treated with cART within 3 months following inclusion in ANRS CO6 Primo Cohort during at least 18 months and cART not modified in the last 3 months
* Controlled on cART: > 90% of VL below 50 cp/mL after initial virological response
* All VL below 50 cp/mL during the previous 12 months
* Most recent CD4 measurement on cART above 500 cells/mm3
* Written and informed consent signed by the person and the investigator (no later than the day of pre-inclusion and prior to any examination realized in the frame of the study (article L1122-1-1 of the Public Health Code)
* Person affiliated or beneficiary of a social security scheme (article L1121-11 of the Public Health Code) (State Medical Aid or AME is not a social security scheme)
* Patient agreeing to participate in the trial according to the defined procedures.

Exclusion Criteria:

* One VL above 1000 cp/mL on or off antitretrovirals after the initial viral control on antiretrovirals was achieved.
* Patient on long-acting injectable HIV treatment
* Patient in whom condom sex use or PrEP use by the partner will be difficult or impossible.
* Woman with a pregnancy project and pregnant woman.
* Patient under guardianship or curatorship.
* History of a clinical AIDS event or cancer.
* Active HCV or HBV infection.
* Any symptoms or laboratory values suggesting a systemic disorder (renal, hepatic, cardiovascular, pulmonary) or other medical conditions, related to HIV or not, which contraindicates the interruption of ARVs.
* Recent SARS-CoV-2 infection and / or associated with a drop in CD4 and / or associated with a resumption of CV in the last 6 months. In this situation, wait until the CD4 has returned to a rate > 500/mm3 and a CV < 50 copies / mL consolidated for > 6 months.
* Affection, disability, resulting from a SARS-CoV-2 infection, regardless of the duration of the SARS-CoV-2 infection.
* Patient participating in another research evaluating other treatments with an exclusion period ongoing at the screening visit.
* Planned absence which could prevent optimal trial participation (vacation abroad, moving, imminent job change ...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with a Plasma HIV-1 RNA (viral load,VL) below 400 copies/mL at 6 months after Treatment interruption (Week 24). | Six months after treatment interruption (Week 24).
  Proportion of subjects with a Plasma HIV-1 RNA below 400 copies/mL on subjects included at 6 months after Treatment interruption.

SECONDARY OUTCOMES:
The acceptation rate of the trial by eligible patients | At inclusion (Day 0)
  Percentage of patients who accept to participate on patients pré-screened and eligible
Proportion of patients with a plasma VL < 50 copies/ml at 3 and 6 months following Analytic Treatment Interruption (ATI) | At 3 months (week 12) and 6 months (week 24) following ATI
  Proportion of patients with a plasma VL < 50 copies/ml at 3 and 6 months following ATI
Evolution of number of CD4 T cells count during ATI and after ART resumption | During all ATI period (from Day 0 to Day 0 ART resumption - maximum 48 weeks) and during ART resumption period (maximum 24 Weeks)
  Measurement of CD4 T cells count at Screening, Day 0, Week 2, Week 4, Week 6, Week 8, Week 12, Week 16, Week 20, Week 24, Week 36, Week 48, Day 0 ART resumption, Week 4 resumption, Week 12 resumption, Week 24 resumption
Evolution of CD4 to CD8 ratio during ATI and after ART resumption | During all ATI period (from Day 0 to Day 0 ART resumption - maximum 48 weeks) and during ART resumption period (maximum 24 Weeks)
  Measurement of CD4 to CD8 at Screening, Day 0, Week 2, Week 4, Week 6, Week 8, Week 12, Week 16, Week 20, Week 24, Week 36, Week 48, Day 0 ART resumption, Week 4 resumption, Week 12 resumption, Week 24 resumption
Evolution of total and integrated HIV DNA and cell-associated HIV RNA transcripts | During ATI period (At Day 0, Week 4, Week 12, Week 24) and during ART resumption period (at Day 0 Resumption, and Week 24 ART Resumption)
  Quantification of total HIV-DNA and integrated HIV-DNA by ultrasensitive techniques (ultrasensitive real-time PCR and Alu PCR) Quantification of intracellular HIV-RNA transcripts by ultrasensitive technique (ultrasensitive qPCR gag).
Evolution of HIV markers in sperm (on 25 participants) | During ATI period (At Day 0, Week 4, Week 12, Week 24) and at Day 0 ART resumption
  Quantification of HIV DNA on semen cells (ultrasensitive technique) and quantification of HIV RNA on seminal fluid (ultrasensitive technique)
Evolution of the levels of inflammation markers during ATI | During ATI period (up to week 24 ATI) and at Day 0 ART resumption
  Physiological parameters levels will be studied (Luminex and Simoa technology): IFNα, TGFβ, IL-7, IL-12, IL-15, IL-18, IP-10, DPPIV, ARNr 16S, I-FABP, citrulline, sCD14, sCD163
Proportion of patients who resumed treatment during the first 6 months of ATI, according to the reasons for resuming | At week 24
  Percentage of resumption, according to the reasons listed in the protocol, before the evaluation of the primary outcome
Pharmacological dosages of antiretrovirals performed during the ATI from frozen samples | At Week 2 and Week 24 of ATI
  Pharmacological dosages of antiretrovirals performed during the ATI at Week 2 and Week 24 of ATI
Proportion of patients reporting at each visit to use condoms | From date of inclusion to the last follow-up visit, up to 72 weeks (average of 1 year).
  Document the emphasis being placed on the impact of access to information on prevention behaviors and the quality of sexual life.
Proportion of patients reporting at each visit to have proposed PrEP at their partners | From date of inclusion to the last follow-up visit, up to 72 weeks (average of 1 year).
  Document the emphasis being placed on the impact of access to information on prevention behaviors and the quality of sexual life.
Proportion of patients satisfied with their participation at the end of the trial | Questionnaire at the end of the study (Week 48 ou Week 24 resumption). Questionnaire at screening (in case of refusal to participate)
  Through statistical analyses of some self-administered questionnaires items (Likert).
  On a Likert scale, a person selects one option among several that reflects how much they agree with a statement. The scale generally consists of five or seven balanced responses that people can choose from.
Evolution of the level of the quality of life between inclusion and the end of the trial | Questionnaire at Day 0, at Week 24 (or resumption of ART) and at the end of the study (Week 48 ou Week 24 resumption). Questionnaire at screening (in case of refusal to participate)
  Through statistical analyses of some self-administered questionnaires items ( SF12.v2 scale for quality of life). The 12-item Short-Form Health Survey is a widely used, generic patient-reported measure of health status that provides summary scores of physical and mental health. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Evolution of the global satisfaction with sexual life between inclusion and the end of the trial | Questionnaire at Day 0, at Week 24 (or resumption of ART) and at the end of the study (Week 48 ou Week 24 resumption). Questionnaire at screening (in case of refusal to participate)
  Through statistical analyses of some self-administered questionnaires items (Likert).
  On a Likert scale, a person selects one option among several that reflects how much they agree with a statement. The scale generally consists of five or seven balanced responses that people can choose from.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile GOUJARD, Principal Investigator — Hôpital Bicêtre, Service de médecine interne et d'immunologie clinique
Locations (30):
- France (30):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Hôtel Dieu, Angers
  - Hôpital Avicenne, Bobigny
  - Hôpital Saint-André, Bordeaux
  - Hôpital PELLEGRIN, Bordeaux
  - Hôpital de la Côte de Nacre, Caen
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Le Bocage, Dijon
  - Hôpital Pierre Zobda-Quitman, Fort de France
  - Hôpital Raymond Poincaré, Garches
  - CHD Vendée, La Roche-sur-Yon
  - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Edouard HERRIOT, Lyon
  - Hôpital Sainte Marguerite, Marseille
  - Hôpital Gui de Chauliac, Montpellier
  - Hôtel Dieu, Nantes
  - Hôpital Carémeau, Nîmes
  - Hôtel Dieu, Paris
  - La Pitié Salpêtrière, Paris
  - Institut Pasteur, Paris
  - Hôpital de l'Hôtel-Dieu, Paris
  - Hôpital Lariboisière, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Tenon, Paris
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Hôpital de Purpan, Toulouse
  - Hôpital Gustave Dron, Tourcoing
  - Hôpital Bretonneau, Tours
  - CHI Villeneuve Saint Georges, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: No